CLINICAL TRIAL: NCT07354789
Title: The Feasibility, Safety and Efficacy of Endoscopic Ultrasound (EUS) Guided Partial Splenic Embolization(PSE): A Cohort Study
Brief Title: The Feasibility, Safety, and Efficacy of EUS-Guided PSE: A Cohort Study
Acronym: EUS; PSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025048
Record Dates: First submitted 2025-12-01; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Cirrhosis; Portal Hypertension; Bleeding
MeSH Terms: conditions — Fibrosis; Hypertension, Portal; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-PSE (Experimental): the patients undergo the PSE via EUS
  Interventions: Procedure: EUS guided PSE

INTERVENTIONS:
Procedure: EUS guided PSE — The patients accepted PSE via EUS

SUMMARY:
Bleeding from esophagogastric varices in patients with liver cirrhosis is often life-threatening. Thrombocytopenia caused by hypersplenism secondary to portal hypertension is an independent risk factor for such gastrointestinal bleeding. Studies have confirmed that partial splenic embolization (PSE) can effectively reduce portal pressure and decrease the risk of rebleeding.

Traditional treatments mainly include total splenectomy and X-ray-guided transarterial partial splenic embolization (X-PSE). Although total splenectomy can completely remove the lesion, its application is limited by issues such as increased risks of postoperative infection, thrombosis, and long-term immune dysfunction. Currently, X-PSE has become the mainstream treatment. This technique involves superselective catheterization of the splenic artery branches using a microcatheter and injecting embolic microspheres to achieve partial splenic embolization, thereby preserving partial splenic function. However, X-PSE relies on radiological intervention techniques and carries risks such as radiation exposure, contrast-induced nephropathy, and non-target embolization (e.g., pancreatic necrosis). Additionally, its ability to locate small arterial branches in the splenic hilum is limited.

Endoscopic ultrasound (EUS) integrates an ultrasound probe at the tip of an endoscope, enabling high-resolution imaging and fine-needle aspiration therapy of the pancreas, gastrointestinal tract, posterior mediastinum, and retroperitoneal structures. With color Doppler functionality, EUS can clearly identify abdominal vessels and their blood flow signals. Since the spleen and splenic vessels are located posterior to the gastric fundus, EUS can clearly visualize the vascular structures of the splenic hilum via a transgastric approach.

Compared to X-PSE, EUS-guided PSE offers the following advantages: a shorter puncture path; avoidance of iodinated contrast agents, making it suitable for patients with iodine allergies or renal insufficiency; no X-ray exposure for patients or operators; the ability to combine treatment for esophagogastric varices in the same procedure, thereby simplifying the process, reducing costs, and shortening hospital stays; and, since there is no arterial puncture site on the body surface, patients do not require prolonged limb immobilization postoperatively, resulting in an overall better healthcare experience.

Current literature and small-sample retrospective studies have reported on this technique, but the included cases are mostly limited to patients with mild liver function impairment, and there is a lack of systematic evaluation of its effect on portal pressure reduction.

The investigators' center integrates the advantages of EUS and X-PSE to perform EUS-guided transgastric puncture for precise injection of embolic materials into the splenic artery branches in patients with liver cirrhosis, gastrointestinal bleeding, and hypersplenism, achieving partial splenic embolization. This study aims to evaluate the safety and efficacy of EUS-guided PSE. The primary endpoint is safety, including the incidence of complications such as intraoperative bleeding, postoperative fever, and abdominal pain scores. Secondary endpoints include efficacy indicators: platelet count, portal pressure gradient, embolization area on CT, incidence of gastrointestinal rebleeding, as well as hospitalization costs and length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years.
2. Diagnosis of liver cirrhosis based on clinical, laboratory, and imaging examinations.
3. Complicated with gastrointestinal bleeding caused by esophagogastric varices.
4. Patients with hypersplenism and thrombocytopenia (platelet count < 100 × 10^9/L).

Exclusion Criteria:

1. Patients who have previously undergone splenectomy, PSE, transjugular intrahepatic portosystemic shunt (TIPS), varicocelectomy, sclerotherapy, or balloon-occluded retrograde transvenous obliteration.
2. Hepatocellular carcinoma or other malignant tumors.
3. Patients with hepatic encephalopathy who are unable to cooperate, or those with liver failure or a Child-Pugh score >13.
4. Patients with allergies to intravenous anesthetics.
5. Patients with unstable vital signs, associated organ dysfunction, active infection, or cardiopulmonary insufficiency, who cannot tolerate endoscopy.
6. Patients who are unable or unwilling to provide informed consent.
7. Uncorrectable coagulation disorders (INR >1.5 and/or fibrinogen <120 mg/dL) or uncorrectable thrombocytopenia (platelet count <20 × 10^9/L).
8. Patients who have used beta-blockers within the past 24 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-12-24 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of intraoperative bleeding | During the EUS-PSE
  The number and rate of patients with intraoperative bleeding.
Postoperative fever | Within one month after the EUS-PSE
  The highest temperature (Celsius degree) of postoperative fever in the patient
Duration of abdominal pain | Within one month after the EUS-PSE
  The duration of the pain (days).
The incidence of recurrent gastrointestinal bleeding | 6 months after the EUS-PSE
  The frequency of esophageal and gastric venous bleeding within six months

SECONDARY OUTCOMES:
Pressure measurements | Before EUS-PSE
  The numerical value of Inferior vena cava pressure (mmHg)、hepatic vein pressure (mmHg)、portal pressure measured pressure (mmHg)、free hepatic venous pressure (mmHg)、wedged hepatic venous pressure (mmHg) via EUS.

OTHER OUTCOMES:
The gender of the patients | At the time of enrollment
  Describe the gender of the patients, including male or female
Etiology of cirrhosis | At the time of enrollment
  Describe the etiology of the cirrhosis
The age of the patients | At the time of enrollment
  The age (years) of the patients.
The number of the platelet | Before EUS-PSE and postoperative follow-up (1 month, 3 months, and 6 months post EUS-PSE )
  The number of the platelet (x 10^9/L)

IPD SHARING:
Plan to Share IPD: Undecided